CLINICAL TRIAL: NCT04682457
Title: Defining the Decline in Endogenous Insulin Secretion in Type 1 Diabetes Diagnosed After 30 Years of Age.
Acronym: DROPLeT
Status: Completed | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2003962
Record Dates: First submitted 2020-12-15; First posted 2020-12-23 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 1; Progression
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Disease Progression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, DNA,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Late Onset: Participants diagnosed with Type 1 diabetes at over 30 years of age.
- 18 to 30: Participants diagnosed with Type 1 diabetes between 18 and 30 years of age

SUMMARY:
The study aims is to find out if people with type 1 diabetes diagnosed in later life (after age 30) have the same rapid loss of insulin secretion (measured using C-peptide) that occurs in younger adults with type 1 diabetes. The investigators will recruit 135 participants aged over 30 years with a clinical diagnosis of type 1 diabetes and diabetes duration ≤100 days. The investigators will also recruit a comparison group of 61 participants aged 18-30 with a clinical diagnosis of type 1 diabetes and diabetes duration ≤100 days. C-peptide will be measured during mixed meal tolerance tests (MMTT) performed at baseline, 6 months and a year.

This study also aims to test a new more practical way of monitoring insulin secretion at home using a finger prick 'blood spot' rather than time consuming tests in a hospital. Finger-prick C-peptide samples will be collected after the MMTT and by the participants at home throughout the year.

DETAILED DESCRIPTION:
The study aims to evaluate progression of type 1 diabetes. Primary analysis will be conducted on those with >=1 diabetes autoantibody positive (GAD, IA2 ZNT8). Sensitivity analysis will be performed by repeating all analysis defining T1D as a) double antibody positivity and b) single antibody positivity combined with a high genetic risk score for T1D (T1DGRS>5th centile of a control population).

Further aims will be to evaluate the utility of dried blood spot testing to detect change in C-peptide and the utility of home test results as a marker of hypoglycaemia and glucose variability.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a clinical diagnosis of Type 1 diabetes within the previous 100 days.
* Aged >30 at the time of Type 1 diabetes diagnosis OR (additional early onset Type 1 diabetes cohort) aged ≥18 and ≤30 at the time of Type 1 diabetes diagnosis.
* Insulin treated at the time of recruitment
* Able and willing to provide informed consent.

Exclusion criteria

* Pregnancy
* Known monogenic diabetes
* Known secondary diabetes (diabetes considered likely due to medication, cystic fibrosis, pancreatitis, pancreatic cancer, pancreatic surgery, hemochromatosis or Cushing's syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recent clinical diagnosis of type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
C-peptide value at a year | 12 months
  12 month (Mixed Meal Tolerance Test) MMTT area under the curve (AUC) C-peptide.
Change in C-peptide over a year | 12 months
  Rate of change of MMTT AUC C-peptide over 12 months assessed at regular study visits

SECONDARY OUTCOMES:
C-peptide value at 12 months | 12 months
  Mean C-peptide at 12 months assessed using MMTT and home blood samples
Glucose variability & hypoglycemia | 12 months
  Glucose variability & hypoglycemia as measured by continuous glucose monitoring (CGM)
Change in dried blood spot C-peptide | 12 months
  Rate of change in home dried blood spot C-peptide over 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Angus Jones, MBBS MRCP, Study Director — NIHR Exeter Clinical Research Facility; Nicholas Thomas, MRCP, Principal Investigator — NIHR Exeter Clinical Research Facility
Locations (1):
- Royal Devon & Exeter NHS Foundation Trust, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thomas NJ, Lynam AL, Hill AV, Weedon MN, Shields BM, Oram RA, McDonald TJ, Hattersley AT, Jones AG. Type 1 diabetes defined by severe insulin deficiency occurs after 30 years of age and is commonly treated as type 2 diabetes. Diabetologia. 2019 Jul;62(7):1167-1172. doi: 10.1007/s00125-019-4863-8. Epub 2019 Apr 10. PMID 30969375